CLINICAL TRIAL: NCT01613963
Title: Observational Study of Visual Outcomes in Retinal Disease
Brief Title: Causes of Visual Loss in Retinal Disease
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Simon Taylor, Senior Lecturer & Consultant Ophthalmic Surgeon, Royal Surrey County Hospital NHS Foundation Trust
Other Study IDs: 12DEV0010
Record Dates: First submitted 2012-05-29; First posted 2012-06-07 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Uveitis; Scleritis
Keywords: Uveitis; Scleritis
MeSH Terms: conditions — Uveitis; Scleritis | interventions — Immunosuppressive Agents; Prednisolone; Azathioprine; Methotrexate; Mycophenolic Acid; Cyclosporine; Infliximab; Adalimumab; Etanercept; Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with ocular inflammation: Patients with ocular inflammation
  Interventions: Drug: Immunosuppressive Agents

INTERVENTIONS:
Drug: Immunosuppressive Agents — Treatment with systemic corticosteroids and/or immunosuppressive agents Treatment with local corticosteroids and other drugs
  Other Names: Prednisolone; Azathioprine; Methotrexate; Mycophenolate mofetil; Cyclosporine A; Infliximab; Adalimumab; Etanercept; Rituximab

SUMMARY:
This is a study of visual outcomes in retinal disease that seeks to identify the causes of visual loss. This data will be used to predict which patients are at risk of losing vision and how they can be better treated.

DETAILED DESCRIPTION:
This is a study of visual outcomes in retinal disease. It is an observational study of patients who have been seen in the retinal clinic, and involves a retrospective casenotes analysis to identify patients who have suffered visual loss and the reason for that visual loss. These data will be analysed to enable the identification of factors that predict visual loss in patients who present earlier in the course of their disease.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of ocular inflammation
* patients with at least 6 months of follow-up

Exclusion Criteria:

* patients without a diagnosis of ocular inflammation
* patients with less than 6 months of follow-up

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ocular inflammation
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Visual acuity at 5 years | 5 years
  Best-corrected visual acuity at 5 years

SECONDARY OUTCOMES:
Visual acuity at 10 years | 10 years
  Best corrected visual acuity at 10 years
Source of referral | Baseline
  Categorised as A&E/GP referral/Optician referral/Tertiary referral
Laterality | Baseline
  Categorised as:
  Right eye/Left eye/Bilateral
Anatomical diagnosis | Baseline
  Cateogorised as:
  Acute anterior uveitis / Chronic anterior uveitis / Fuchs heterochromic cyclitis / Intermediate uveitis / Pars planitis / Posterior Uveitis / Panuveitis / Episcleritis / Scleritis
Aetiological diagnosis | Baseline
  Diagnosed as:
  Viral / Bacterial / Fungal / Parasitic / Inflammatory / Malignant
Associated systemic disease | Baseline
  Any associated systemic disease, e.g. HLA-B27 associated disease, Behcet's disease, multiple sclerosis, Vogt-Koyanagi-Harada syndrome, rheumatoid arthritis, collagen vascular disease, tuberculosis, granulomatosis with polyangiitis
Complications of disease and causes of visual loss at 5 years | 5 years
  Categorised into:
  Corneal clarity problems / cataract / vitreous debris / retinal detachment / cystoid macular edema / retinal pigment epithelium atrophy / macular scarring / epiretinal membrane / macular hole / steroid response / glaucoma / other optic neuropathy / hypotony & phthisis / other
Complications of disease and causes of visual loss at 10 years | 10 years
  Categorised into:
  Corneal clarity problems / cataract / vitreous debris / retinal detachment / cystoid macular edema / retinal pigment epithelium atrophy / macular scarring / epiretinal membrane / macular hole / steroid response / glaucoma / other optic neuropathy / hypotony & phthisis / other
Complications of disease and causes of visual loss | Up to 10 years
  Categorised into:
  Corneal clarity problems / cataract / vitreous debris / retinal detachment / cystoid macular edema / retinal pigment epithelium atrophy / macular scarring / epiretinal membrane / macular hole / steroid response / glaucoma / other optic neuropathy / hypotony & phthisis / other
Treatment measures employed | Up to 10 years
  Categorised into:
  Topical treatment / periocular steroid / intraocular steroid / intraocular other agent / Glaucoma treatment / systemic immunosuppressive agents
Complications of disease and treatment | Up to 10 years
  Categorised into:
  1. Local complications: Raised intraocular pressure / cataract / endophthalmitis / other
  2. Systemic complications: Diabetes / hypertension / cholesterol / liver function / bone density loss / other
Surgical procedures | Up to 10 years
  List and dates of any intraocular surgery performed during the study
Burden of disease - appointments | Up to 10 years
  Number of outpatient appointments over the course of the study
Burden of disease - outpatient procedures | Up to 10 years
  Number of outpatient procedures over the course of the study
Burden of disease - inpatient procedures | Up to 10 years
  Number of inpatient procedures over the course of the study
Blind registration | Up to 10 years
  Year of any registration as partially sighted or blind

CONTACTS AND LOCATIONS:
Overall Officials: Simon RJ Taylor, PhD FRCOphth, Principal Investigator — Royal Surrey County Hospital NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Moorfields Eye Hospital, London, London
  - Royal Surrey County Hospital, Guildford, UK